CLINICAL TRIAL: NCT01048255
Title: A Phase 2, Randomized, Double-blind,Placebo-controlled Study of VX-765 in Subjects With Treatment-resistant Partial Epilepsy
Brief Title: Study of VX-765 in Subjects With Treatment-resistant Partial Epilepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX09-765-401
Record Dates: First submitted 2010-01-08; First posted 2010-01-13 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2013-12

CONDITIONS: Partial Epilepsy
MeSH Terms: conditions — Epilepsies, Partial | interventions — belnacasan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- VX-765 (Experimental)
  Interventions: Drug: VX-765

INTERVENTIONS:
Drug: VX-765 — 300mg Oral Tablet, 900mg TID

SUMMARY:
The purpose of this study is to determine the safety, tolerability, and efficacy of VX-765 in subjects with Treatment-resistant Partial Epilepsy

ELIGIBILITY:
Inclusion Criteria:

* Subjects that are male or female aged 18 to 64 years (inclusive) with a body mass index between 18 and 35 (kg/m2)
* Subjects must have a diagnosis and history of treatment resistant partial onset seizures for which they are taking 1 to 4 concomitant antiepileptic drugs (AED). Treatment resistance is defined as failure to achieve seizure freedom despite adequate use of 2 different AEDs. All AED doses must remain stable for 4 weeks prior to the Screening Visit and throughout the entire study
* Subjects must have had at least 1 electroencephalogram (EEG) consistent with partial epilepsy and a brain magnetic resource imaging (MRI) or computed tomography (CT) scan within 5 years of Screening Visit negative for other confounding conditions
* Subjects must have had at least 6 observable partial seizures in 6 weeks prior to randomization, with at least 1 seizure per week during 3 of the 6 weeks within the Baseline Period
* Subjects who are male or female must agree to use acceptable contraceptive methods as defined in the protocol
* Subjects who are in otherwise good health

Exclusion Criteria:

* Subjects with a history of non-epileptic transient alterations in consciousness
* Subjects who have a history of status epilepticus in the past 12 months
* Subjects whose seizure frequency cannot be quantified
* Subjects who have significant medical illness including kidney, liver, pulmonary or gastrointestinal disease; or unstable or poorly controlled conditions
* Subjects who have clinically significant psychiatric illness
* Subjects with a positive drug screen (excluding any allowed prescribed medications) and history of alcoholism or drug addiction within past 2 years
* Males subjects that have a female partner of childbearing potential who do not agree to use medically approved methods of birth control
* Male subjects that have a female partner who is pregnant, nursing, or is planning to become pregnant during the study period, or within 90 days of the last dose of study drug
* Female subjects who are pregnant or lactating, or who are of reproductive potential who do not agree to use medically approved birth-control methods
* Subjects with a current or prior history of illness precluding them from immunomodulatory therapy (e.g. history of recurrent infections)
* Subjects with active hepatitis B, hepatitis C, or human immunodeficiency virus (HIV)
* Subjects who have participated in any other clinical trials involving an investigational product or device and have received the last dose of study drug within 45 days or 5 half-lives of the Screening Visit

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2010-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability (vital sign assessments, physical and neurological examinations, laboratory assessments, and adverse events) | 18 weeks

SECONDARY OUTCOMES:
Percent reduction in seizure frequency | 6 weeks
Percent of subjects with 50% or greater reduction in seizure frequency | 6 weeks
Percent of subjects that become seizure free | 2 weeks
Percent of subjects who discontinue study drug treatment | 6 weeks
Plasma levels of study drug and other concomitant antiepileptic drugs | 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chris Wright, MD, PhD, Study Director — Vertex Pharmaceuticals Incorporated
Locations (12):
- United States (12):
  - Arkansas, Little Rock, Arkansas
  - California, Newport Beach, California
  - Florida, Miami, Florida
  - Florida, Sarasota, Florida
  - Illinois, Chicago, Illinois
  - Maryland, Baltimore, Maryland
  - Maryland, Bethesda, Maryland
  - Missouri, Chesterfield, Missouri
  - New Jersey, Hackensack, New Jersey
  - New York, New York, New York
  - Pennsylvania, Philidelphia, Pennsylvania
  - Virginia, Charlottesville, Virginia

REFERENCES:
- [Derived] Panebianco M, Walker L, Marson AG. Immunomodulatory interventions for focal epilepsy. Cochrane Database Syst Rev. 2023 Oct 16;10(10):CD009945. doi: 10.1002/14651858.CD009945.pub3. PMID 37842826